CLINICAL TRIAL: NCT05628766
Title: The Role of Thiol/Disulphide Homeostasis in Unexplained Primary Infertile Patients
Brief Title: Thiol/Disulphide Homeostasis in Unexplained Infertility
Status: Completed | Type: Observational
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Serif Aksin, associate professor, Siirt University
Other Study IDs: SiirtUNIVERSI
Record Dates: First submitted 2022-11-07; First posted 2022-11-29 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Oxidative Stress; Infertility; Antioxidative Stress
MeSH Terms: conditions — Infertility | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women diagnosed with primary infertility (n:41): Women which followed up with infertility of unknown cause.
  Interventions: Other: complete blood count
- Control group ( n:41): Healthy women who are not infertile
  Interventions: Other: complete blood count

INTERVENTIONS:
Other: complete blood count — Thiol/disulphide levels in the blood will be checked by taking complete blood count

SUMMARY:
The aim in this study is to determine whether there is a relationship between Thiol / Disulphide levels in primary infertile patients and comparing them with infertile patients and the control group. For this purpose, 41 women followed up with the diagnosis of primary infertility in Siirt Training and Research Hospital between November 2022 and January 2023 will be included in the study. The same number of (n:41) non-infertile control women will be included. Age, pregnancy history and medical history of both groups will be recorded. FSH, LH, E2, TSH, and prolactin levels taken routinely in these patients will be examined. Thiol/disulphide levels in the blood will be checked by taking whole blood from these patients. In the light of the information thus obtained, the investigator plan to determine whether there is a relationship between oxidant/antioxidant balance in primary infertile patients.

DETAILED DESCRIPTION:
Reactive oxygen species (ROS) are products of normal cellular metabolism and consist of oxygen ions, free radicals and peroxides. Adding an electron to oxygen creates the superoxide anion radical, which can then be converted to a hydroxyl radical, peroxyl radical, or hydrogen peroxide. Free radicals try to participate in chemical reactions that free themselves of their unpaired electrons and result in oxidation. Natural antioxidants found in the body include catalase, glutathione peroxidase, superoxide dismutase and glutathione reductase, vitamins C and E, ferritin, and transferrin. Other lifestyle factors such as smoking, diet, illness, pollution, stress, alcohol, and allergies also contribute to increased levels of free radicals, suggesting that these factors have a negative impact on female fertility, potentially through the formation of excessive oxidative stress.

Excessive accumulation of ROS can damage cells, proteins, DNA and lipids; therefore, ROS levels are regulated by antioxidant mechanisms in the organism. A shift in the direction of ROS in this balance is called oxidative stress (OS). ROS produced in the follicle have important roles in folliculogenesis and ovulation. Granulosa cells produce antioxidants to protect oocytes from the harmful effects of excess ROS. OS has been implicated as an etiopathogenetic factor in female infertility. The number of studies examining the role of OS in the etiopathogenesis of infertility has increased in recent years, and it has been suggested that increased OS and/or decreased antioxidant defense mechanisms may contribute to infertility-related conditions.

One of the defense mechanisms against OS in humans is the thiol redox reaction. The thiol consists of a sulfhydryl group, and under OS conditions these functional groups form reversible disulfide bridges. These bonds bring about functional and structural changes in proteins. Disulfide bonds are reduced to thiol groups through antioxidant mechanisms, thereby providing thiol/disulfide homeostasis. Thus, disulfide bridges are thought to be a marker of OS, while thiols are suggested to be members of the antioxidant system. Only one side of this equilibrium has been measured by Ellman (1979), whereas in recent years both sides of the thiol/disulfide equilibrium can be measured by the Erel and Neselioğlu assay method, allowing a full assessment of the thiol/disulfide status.

Dynamic thiol/disulfide homeostasis, a recently identified marker of OS, is thought to have critical roles in pathological processes in various vital processes such as folliculogenesis and ovulation.

n the literature review, there are studies investigating the relationship between infertility and oxidant/antioxidants. However, measurements require measuring a large number of parameters and many separate biomarkers. The thiol/disulfide balance is beneficial in terms of showing the oxidant/antioxidant balance in total. It was not possible to measure this balance simultaneously on both sides in the method measuring the thiol/disulfide balance by Newman in 1979. In recent years, it has become possible to measure the serum Thiol/disulfide balance bilaterally with the automatic spectrophotometric method described by Erel and Neşelioğlu. This study aims to investigate whether there is a relationship by measuring the Total oxidant/antioxidant load with the Thiol/disulfide method in patients with unexplained infertility, to investigate the relationship between thiol/disulfide homeostasis and impaired ovulation and fertility, and to analyze the potential pathogenetic mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary infertility
* Patients between the age of 18-35

Exclusion Criteria:

* Active hypertension
* Chronic liver or kidney failure history
* Coronary artery disease
* Acute infection (within 14 days)
* Any chronic inflammatory disease
* Presence of autoimmune disease
* Known malignancy
* Inflammatory bowel disease
* Hormonal contraception
* Smoking
* alcohol use
* Drug use
* Patients with tubal infertility
* Partner with abnormal spermiogram

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Women between the age of 18-35 diagnosed with infertility of unknown cause.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Measuring the total oxidant/antioxidant load with the Thiol/disulfide method in patients with unexplained infertility | "through study completion, an average of 4 months
  To determine whether there is a relationship between oxidant/ antioxidant balance in primary infertile patients by looking at Thiol/disulphide blood levels in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Şerif Aksin, assoc.Prof, Study Director — Siirt University Medical Faculty Obstetrics and Gynecology Departmant
Locations (1):
- Siirt Üniversity Medical Faculty, Siirt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No